CLINICAL TRIAL: NCT03567993
Title: mHealth Messaging to Motivate Quitline Use and Quitting (M2Q2): RCT in Rural Vietnam
Brief Title: mHealth Messaging to Motivate Quitline Use Quitting
Acronym: M2Q2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Institute of Population, Health and Development, Vietnam (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Rajani Sadasivam, Associate Professor, Population and Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00012953; R01TW010647 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Tobacco Use Cessation
Keywords: mhealth; Tobacco cessation; Vietnam; Smoking cessation
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison (Active Comparator): The comparison condition is designed as a minimal intervention, and allows for blinding of the patients to randomization group.
  Interventions: Behavioral: Comparison
- Intervention (Experimental): The intervention is designed to encourage and remind smokers of the availability of the Quitline services. In addition to the one-way motivational messages, the investigators will use two-way assessments. Two-way automated texting is the ability to push out a question, have the user respond with a brief, numeric or one-word answer, and based on that answer, provide immediate feedback. The goal of these brief assessments is two-fold: 1) to assess behavior (abstinence) and motivation to use services, and 2) to return feedback tailored to each individual smoker based on the answers of the user.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Comparison — Participants randomized to the comparison arm will receive twice-monthly abstinence assessments from the text messaging system, with no motivational feedback. Those in the comparison arm are neither offered nor encouraged to participate in the intervention.
  Arms: Comparison
Behavioral: Intervention — Participants randomized to the intervention arm will receive:
  1. Motivational Messages
  2. Abstinence and Motivation to Use Services Assessments
  3. Encouragement to access the Quitline
  4. Encouragement to use Nicotine Replacement Therapy (NRT)
  5. Provision of NRT, if requested
  Intervention subjects are encouraged to access the Quitline and use NRT. However, these are not mandatory components of the intervention and subjects can choose if they would like to engage with the Quitline or use NRT.
  Other Names: mHealth Intervention
  Arms: Intervention

SUMMARY:
The mHealth Messaging to Motivate Quitline Use and Quitting, or "M2Q2" study, is a collaborative research project for a mobile health intervention designed to motivate smoking cessation and encourage access to counseling. The study is for men and women smokers in Vietnam's Red River Delta region who are 18 years of age or older.

The primary hypothesis is that smokers in the M2Q2 intervention will have higher rates of smoking cessation, compared with the comparison group.

DETAILED DESCRIPTION:
The specific aims of the M2Q2 study are:

Aim 1: In collaboration with the Institute of Population, Health, and Development (PHAD) in Vietnam, adapt a current, effective messaging system to Vietnam. The messaging system will:

1. Motivate smokers to quit smoking, using tailored messages adapted to be culturally relevant.
2. Encourage smokers to accept counseling services from the Quitline, and take advantage of nicotine replacement therapy (NRT) that will be provided by the Quitline to those willing to quit.

Aim 2: To engage with the Quitline, providing additional training in tobacco cessation counseling for those ready to quit, and motivational interventions for those not yet ready to quit.

Aim 3: To evaluate the impact of the messaging system on: access to the Quitline, use of nicotine replacement therapy, increase in self-efficacy, and six-month biochemically verified smoking cessation.

The study will be conducted in the Red River Delta Region, an agriculturally rich and densely populated area in northern Vietnam. Four communes (Viet Hung, Binh Minh, Tan Viet and Bach Sam) located in four different districts in the Hung Yen province will be included in the M2Q2 study, based on their general representativeness to the rural northern Vietnamese population and because the investigators have developed infrastructure to support technology-assisted behavioral interventions through community health centers (CHCs) in these communes. Each of the selected communes satisfy the following criteria: (1) have a community health center with a medical doctor; (2) are not currently participating in other studies for smoking cessation; and (3) have a minimum geographic separation of 12 kilometers (7 miles) from all other study communes to minimize possible contamination.

Recruitment and retention of study participants will be conducted by both CHC staff and community health workers. The investigators will recruit men and women, and plan for recruiting 15% women. The investigators will plan to recruit smokers regardless of their readiness to quit. Participants will not be compensated, other than being provided a cellphone if they currently do not own one.

The duration of an individual subject's participation in the study is 6 months (baseline survey, texting system, quitline data, and the 6-month follow-up survey). The duration anticipated to enroll all study subjects is 2 years, 2 months. The estimated date for the investigators to complete this study with primary analyses is the middle of year 5.

The main dependent variable is patient tobacco cessation rate (quit rate) at six months. The investigators will biochemically verify smoking status at baseline and at six months. The secondary outcome measure is self-efficacy. The investigators will administer an 12-item questionnaire (SEQ-12) to measure self-efficacy at baseline and at six months.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Resident of a selected commune.
3. Be a current smoker.
4. Be able to receive texts and read text (literate).
5. Not be cognitively impaired (as assessed by study staff).
6. Not have helped develop messages used in the intervention.
7. Not be a family member of another participant in the study.

Exclusion Criteria:

1. <18 years of age.
2. Cognitively impaired (as assessed by study staff).
3. Pregnant.
4. Prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajani S Sadasivam, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Institute of Population, Health, and Development (PHAD), Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.

REFERENCES:
- [Derived] Larkin C, Wijesundara J, Nguyen HL, Ha DA, Vuong A, Nguyen CK, Amante D, Ngo CQ, Phan PT, Pham QTL, Nguyen BN, Nguyen ATP, Nguyen PTT, Person S, Allison JJ, Houston TK, Sadasivam R. mHealth Messaging to Motivate Quitline Use and Quitting: Protocol for a Community-Based Randomized Controlled Trial in Rural Vietnam. JMIR Res Protoc. 2021 Oct 7;10(10):e30947. doi: 10.2196/30947. PMID 34617915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred over a 22-month period, from November 23, 2018, through October 7, 2020.
Pre-assignment Details: During monthly recruitment events, study staff screened interested individuals for eligibility, consented, and enrolled eligible individuals in the study. Enrolled participants completed a baseline survey before randomization. No participants were excluded between enrollment and assignment to study arms.
Groups:
- Intervention: The intervention is designed to encourage and remind smokers of the availability of the Quitline services. In addition to the one-way motivational messages, the investigators will use two-way assessments. Two-way automated texting is the ability to push out a question, have the user respond with a brief, numeric or one-word answer, and based on that answer, provide immediate feedback. The goal of these brief assessments is two-fold: 1) to assess behavior (abstinence) and motivation to use services, and 2) to return feedback tailored to each individual smoker based on the answers of the user.
  Intervention: Participants randomized to the intervention arm will receive:
  1. Motivational Messages
  2. Abstinence and Motivation to Use Services Assessments
  3. Encouragement to access the Quitline
  4. Encouragement to use Nicotine Replacement Therapy (NRT)
  5. Provision of NRT, if requested
  Intervention subjects are encouraged to access the Quitline and use NRT. However, these are not mandatory components of the intervention and subjects can choose if they would like to engage with the Quitline or use NRT.
Period: Overall Study
Arm/Group | Comparison | Intervention
Started | 378 | 372
Completed | 372 | 369
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One comparison participant did not complete the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparison | Intervention | Total
Number analyzed (Participants) | 377 | 372 | 749
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 364 | 364 | 728
  >=65 years | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.6) | 42.7 (12.5) | 42.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 377 | 372 | 749
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 377 | 372 | 749
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 377 | 372 | 749
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 377 | 372 | 749
Baseline Smoking Self-Efficacy (SEQ-12) Questionnaire [Mean (Standard Deviation); unit: Scores on a Scale] — The Smoking Self-Efficacy Questionnaire (SEQ-12) measures the self-reported confidence of current and former smokers in their ability to abstain from smoking in high-risk situations (e.g., when facing internal stimuli (e.g., feeling depressed) and external stimuli (e.g., being with smokers)). The SEQ-12 consists of 12 items; each item is rated on a 5-point Likert scale (1=not at all sure, 2=not very sure, 3=more or less sure, 4=fairly sure, and 5=absolutely sure). SEQ-12 scores range from 12 to 60, with higher scores indicating greater self-efficacy. Items are summed to compute total score.
  Scores on a Scale | 33 (9.9) | 32 (9.9) | 32.8 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Participant Tobacco Cessation Rate (Quit Rate) at 6 Months
Description: 7 day point prevalence cessation per self-report with additional carbon monoxide monitor verification for those who report cessation.
Time Frame: At 6 months post-randomization
Population: The number of participants analyzed did not differ from the number of participants assigned to the arm or comparison group.
Measure: Number; unit: proportion of participants
Arm/Group | Comparison | Intervention
Number analyzed (Participants) | 372 | 369
proportion of participants | .50 | .52

2. Secondary Outcome: Change in Self-efficacy Scores Using the Self Efficacy Questionnaire (SEQ-12)
Description: Study team will administer the Self Efficacy Questionnaire (SEQ-12), an 12-item questionnaire to measure self-reported confidence of current and former smokers in their ability to abstain from smoking in high-risk situations (e.g., when facing internal stimuli (e.g., feeling depressed) and external stimuli (e.g., being with smokers)). The SEQ-12 consists of 12 items; each item is rated on a 5-point Likert scale (1=not at all sure, 2=not very sure, 3=more or less sure, 4=fairly sure, and 5=absolutely sure). SEQ-12 scores range from 12 to 60, with higher scores indicating greater self-efficacy. Individual items are summed to compute the total score. The outcome will measure the change in SEQ-12 scores from baseline to 6 months post-randomization.
Time Frame: From randomization to 6 months post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SEQ-12 scores
Arm/Group | Comparison | Intervention
Number analyzed (Participants) | 372 | 369
SEQ-12 scores | 43 (10.2) | 43 (10.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 6 months.
Description: The study used the clinicaltrials.gov definition of adverse events and serious adverse events.
Arm/Group | Comparison | Intervention
All-Cause Mortality (participants affected / at risk) | 1/378 | 1/372
Serious Adverse Events (participants affected / at risk) | 1/378 | 1/372
Other Adverse Events (participants affected / at risk) | 0/378 | 0/372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparison (N=378) | Intervention (N=372)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The participant had an underlying disease (COPD) and died of acute bronchospasm on 10/15/2019. This event was unrelated to the study.
Death (Cardiac disorders) | 0 (0) | 1 (1) — The participant died at home at 13:00 on 12/16/2019 due to a stroke. This event was unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03567993/Prot_SAP_000.pdf